CLINICAL TRIAL: NCT01110174
Title: Assessing Response to Neoadjuvant Chemotherapy With Dedicated Breast High Definition PET/CT, Serum Glycomic Markers and Tissue Muc-1 Isoforms
Brief Title: Assessing Response to Neoadjuvant Chemotherapy With HD PET/CT, Serum Glycomic Markers and Tissue Muc-1 Isoforms
Acronym: ENIGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 216529; CCSO 010
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HD PET/CT (Experimental): utilization of PET/CT for diagnostic of breast cancer progression.
  Interventions: Diagnostic Test: HD PET/CT

INTERVENTIONS:
Diagnostic Test: HD PET/CT — imaging

SUMMARY:
A pilot study of adult (≥ 18 years) women with stage II-III breast cancer who will receive preoperative chemotherapy prior to mastectomy. Patients will have real-time serum glycan profiling, expression of tissue MUC 1 oncoprotein isoforms to predict neoadjuvant chemotherapy response and additional mammography and HD PET/CT examinations to assess response. The investigators hypothesize that a functional tumor assessment utilizing high-definition positron emission tomography/computed tomography (HD PET/CT), real-time serum glycan profiling, and expression of tissue MUC 1 oncoprotein isoforms will predict neoadjuvant chemotherapy response in breast cancer patients.

DETAILED DESCRIPTION:
This is a non-randomized clinical trial pilot study. Consenting adult (≥ 18 years) women with stage II-III breast cancer undergoing will receive neoadjuvant chemotherapy with a standard ACT regimen prior to mastectomy. Prior to beginning chemotherapy, patients will receive a baseline mammogram, breast HD PET/CT, and blood draw. Not more than 7 days prior to the second cycle of chemotherapy, patients will have both HD PET/CT and diagnostic mammography images taken to assess early response to treatment. Patients will have two additional mammography and HD PET/CT examinations: one after the first cycle of chemotherapy, and another upon completion of the last cycle of chemotherapy but before mastectomy. The investigators will collect data on the size (maximum diameter, estimated volume) and 18FDG uptake (SUV) of the known primary breast cancer on HD PET/CT. Blood will be sampled from patients at 12 separate time points during the study for glycan analysis. At least 3 ml will be taken with each blood draw. The first blood draw will be taken when the patient agrees to enroll in the study. The second blood draw will be taken prior to the first cycle of chemotherapy. Thereafter, blood will be drawn for serum glycan analysis after each cycle of chemotherapy is completed. After the patient undergoes mastectomy, tissue will be collected for MUC-1 assay and two additional blood draws will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign informed consent to participate in the study.
* Patient must be ≥ 18 years of age.
* Histologic diagnosis of invasive breast cancer(ductal or lobular)
* Stage II or III breast cancer and considered a candidate for curative mastectomy.
* Selected mastectomy for surgical option of treatment.
* Patient must agree to receive standard or dose-dense adriamycin, cyclophosphamide, and taxane-based chemotherapy given preoperatively.
* Patient must have the following preoperative laboratory values confirmed within 28 days prior to registration: Creatinine ≤ 1.5 times ULN. Platelets ≥ 90,000/mm3. White blood count ≥ 1,500/mm3. PT/PTT ≤ the institution ULN. Patients of child-bearing potential must have a negative urine or serum pregnancy test.
* If a patient is a cancer survivor, the patient must have undergone potentially curative therapy for all prior malignancies, with no evidence of prior malignancy for at least 5 years (except for effectively treated basal cell or squamous cell carcinoma of the skin, or carcinoma-in-situ of the cervix treated by surgery alone).
* The primary breast tumor must be detectable by mammogram at the time of diagnosis
* Estimated cardiac ejection fraction ≥ 50% by echocardiogram or MUGA
* ECOG performance status 0-1.

Exclusion Criteria:

* Non-invasive breast cancer, benign breast disease, or tumor histology other than stage II or stage III invasive ductal carcinoma, invasive lobular carcinoma, or mixed ductal and lobular carcinoma.
* The patient has known distant metastatic disease.
* The patient wishes to pursue breast conservation.
* The patient is male.
* The patient is receiving preoperative chemotherapy other than adriamycin, cyclophosphamide, and a taxane (ACT) in standard or dose-dense fashion.
* The patient is pregnant or breast feeding.
* The primary tumor is not visualized by mammogram at the time of diagnosis.
* The patient's estimated cardiac ejection fraction is <50% by echocardiogram or MUGA.
* The patient has a documented intravenous contrast allergy or iodine allergy.
* Her-2/neu positive patients by IHC or FISH who receive trastuzumab neoadjuvantly; patients who are Her-2/neu positive but elect not to receive trastuzumab neoadjuvantly are still eligible for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Martinez, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HD PET/CT
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HD PET/CT
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
  Between 18 and 65 years | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
  >=65 years | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
  Male | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
Region of Enrollment [Number; unit: participants]
  United States | NA — PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data

OUTCOME MEASURES:

1. Primary Outcome: Assess the Ability of the HD PET/CT to Predict Final Histopathologic NAC Response.
Description: Patients will have a HD PET/CT at baseline and another after the first cycle of NAC and upon completion.The goal is to distinguish NAC responders from non-responders and to accurately identify the size and extent of residual disease.
Time Frame: After the first cycle of Neoadjuvant chemotherapy (NAC)
Population: PI has left the institution, all efforts to locate PI and obtain this information have been exhausted and there is no access to this data
Arm/Group | HD PET/CT
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlate Serum Circulating BCa-related Glycan Profiles With Radiographic and Histopathologic Assessments of NAC Response.
Time Frame: Baseline, during and after chemotherapy
Population: PI has left institution, all efforts to locate secondary outcome measure data have been exhausted and there is no longer access to this data.
Arm/Group | HD PET/CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HD PET/CT
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Dr. Martinez, left UC Davis in 2013 and Dr. Bold was listed as PI. No new participants were enrolled under Dr. Bold, and he does not have access to the data. UC Davis does not have any means of contacting Dr. Martinez pursuant to results entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes